CLINICAL TRIAL: NCT07202962
Title: Study of Prevalence of Inappropriate Prescriptions in Hospitalized Elderly Patients According to STOPP&Amp;START Criteria (Screening Tools of Older Person Prescriptions and Screening Tool to Alert to Right Treatment) - SPIna Protocol
Brief Title: Prevalence of Inappropriate Prescriptions and Omitted Therapies in Hospitalized Elderly: STOPP/START Criteria Analysis
Acronym: SPIna
Status: Completed | Type: Observational
Sponsor: Regione del Veneto - AULSS n. 7 Pedemontana (Other)
Responsible Party: Principal Investigator, Luca Pellizzari, Director of Geriatrics, Regione del Veneto - AULSS n. 7 Pedemontana
Other Study IDs: 1239
Record Dates: First submitted 2025-02-27; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2024-12

CONDITIONS: Polypharmacy (People Under Treatment With 5 or More Drugs); Elderly (People Aged 65 or More); Deprescribing; Hospitalization
Keywords: polypharmacotherapy; interactions; elderly people; STOPP&START CRITERIES; DEPRESCRIBING
MeSH Terms: interventions — Medication Review; Deprescriptions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: medication review and deprescribing — The study protocol includes the following assessments:
  * T0: first data collection upon admission to the ward;
  * T1 assessment: pharmacological review at discharge. Subjects who meet all study eligibility criteria will come consecutively enrolled in the study during admission to the department (T0).
  By consulting the electronic health record, interviewing patients and family members and personal documentation, the following data will be collected:
  * Remote and immediate pathological history;
  * Family and social history;
  * Home therapy;
  * BRIEF-MPI. Home therapy and therapy suggested at discharge will be compared with the STOPPandSTART criteria to evaluate the prevalence of potential therapies inappropriate and to study possible interactions and contraindications pharmacological and for reporting possible adverse reactions to drugs. The prevalence and possible prevalence of each individual STOPPandSTART criterion will be assessed association with other variables of interest.

SUMMARY:
Evaluate the prevalence of potentially inappropriate prescriptions (PIPs) and potential omitted prescriptions (PPOs) in elderly patient upon admission to the acute geriatric department, based on adherence or non-adherence to the recommendations specified in STOPP and START criteria.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients (aged >75 years) admitted to the Geriatrics Department at Santorso, Alto Vicentino Hospital.
* Currently undergoing pharmacological treatment at the time of admission.

Exclusion Criteria:

• Patients placed in palliative therapy upon admission to the department due to incurability of the underlying pathologies

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients aged over 75 years on polypharmacotherapy, hospitalized for acute conditions in the Geriatrics Department of AULSS 7 Pedemontana Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-07-17 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of Potentially Inappropriate Prescriptions (PIP) (%) | Data collected at time Day 0 is analyzed by day 4. Data collected at time Day 1 is analyzed by day 4
  Percentage of elderly patients with at least one potentially inappropriate prescription identified at hospital admission (day 0) and at discharge (day 1) in the acute geriatric ward, based on the STOPP criteria. The measurement is performed by comparing the patient's medication regimen with the recommendations provided in the STOPP criteria.
Prevalence of Potentially Omitted Prescriptions (PPO) (%) | Data collected at time Day 0 is analyzed by day 4. Data collected at time Day 1 is analyzed by day 4
  Percentage of elderly patients with at least one potentially omitted prescription identified at hospital admission (day 0) and at discharge (day 1) in the acute geriatric ward, based on the START criteria. The measurement is based on the absence of indicated medications according to the START criteria recommendations.

SECONDARY OUTCOMES:
Prevalence of Pharmacological Interactions (%) | Data collected at time Day 0 is analyzed by day 4. Data collected at time Day 1 is analyzed by day 4
  Percentage of patients with at least one clinically significant drug-drug interaction identified through analysis of the medication regimen using standard drug interaction checkers. Assessed at admission and discharge.
Post-Discharge Destination (Binary Variable) | Data collected at time Day 0 is analyzed by day 4.
  Discharge destination classified as a binary variable (e.g., Home vs. Institutional care). Each category is analyzed separately.
Presence of Geriatric Syndromes (Yes/No) | Data collected at time Day 0 is analyzed by day 4.
  Presence of specific geriatric syndromes (e.g., delirium, falls, incontinence, pressure ulcers, etc.) assessed as separate binary variables (Yes/No) for each syndrome, based on clinical records and standardized assessment tools.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Pellizzari Dr. Pellizzari, DR, Principal Investigator — Regione del Veneto - AULSS n. 7 Pedemontana
Locations (1):
- Regione del Veneto - AULSS n. 7 Pedemontana, Santorso, Vicenza, Italy